CLINICAL TRIAL: NCT01203215
Title: Evaluating Self-Help Programs for Exercise Adoption and Maintenance in Women
Brief Title: Examining Two Print-based Exercise Interventions for Women
Acronym: WWP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: The Miriam Hospital (Other)
Responsible Party: Melissa A Napolitano, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RWJF044224
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2010-09

CONDITIONS: Physical Activity Behavior
Keywords: exercise; physical activity; women; community
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- JumpStart (Experimental)
  Interventions: Behavioral: 2 print based physical activity interventions
- Choose to Move (Experimental)
  Interventions: Behavioral: 2 print based physical activity interventions
- Wellness (Active Comparator)
  Interventions: Behavioral: 2 print based physical activity interventions

INTERVENTIONS:
Behavioral: 2 print based physical activity interventions — physical activity promotion

SUMMARY:
Print-based interventions, specifically interventions that are theoretically-based have been shown to be effective for individuals. These types of interventions are of particular importance for those individuals who, due to transportation, work, family, social, or financial demands have difficulty participating in face-to-face programs. Therefore, we decided to test 2 such print based programs for women.

DETAILED DESCRIPTION:
We conducted a randomized controlled trial in which participants were randomly assigned to one of three groups: (1) Choose to Move (CTM), a gender-targeted intervention (2) Jumpstart, a motivationally-tailored print-based intervention, or (3) Wellness contact control group. Objective and self-report measures of physical activity and psychosocial mediators of change were assessed at 3 months to evaluate the efficacy of the programs and maintenance of these programs will be conducted by examining a 9 month follow-up phase. This design allows a direct comparison between two print-based physical activity self-help programs. The use of non face-to-face interventions is critical to reach the large numbers of women in United States who are not physically active. Tailored print materials (i.e., Jumpstart) will enable participants to have information that is matched to their level of motivation, and thus might be expected to be more efficacious than a standard self-help intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy women
* sedentary

Exclusion Criteria:

* participating in > 90 minutes of purposeful physical activity (e.g., walking, cycling).
* medical problems that could potentially impede or exacerbated by physical activity
* history of coronary heart disease
* myocardial infraction
* symptoms of angina
* stroke
* diabetes
* osteoporosis
* osteoarthritis
* severe orthopedic problems.
* a planned move from the area within the next year
* current or planned pregnancy
* hospitalization for a psychiatric disorder within the last 3 years
* current suicidal or psychotic episodes
* currently using certain prescription medication such as beta blockers for hypertension

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2002-06; Primary Completion 2005-06 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Physical activity | 3 months

SECONDARY OUTCOMES:
physical activity | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Napolitano MA, Whiteley JA, Papandonatos G, Dutton G, Farrell NC, Albrecht A, Bock B, Bazzarre T, Sciamanna C, Dunn AL, Marcus BH. Outcomes from the women's wellness project: a community-focused physical activity trial for women. Prev Med. 2006 Dec;43(6):447-53. doi: 10.1016/j.ypmed.2006.06.011. Epub 2006 Aug 17. PMID 16919322
- [Result] McAndrew LM, Napolitano MA, Albrecht A, Farrell NC, Marcus BH, Whiteley JA. When, why and for whom there is a relationship between physical activity and menopause symptoms. Maturitas. 2009 Oct 20;64(2):119-25. doi: 10.1016/j.maturitas.2009.08.009. Epub 2009 Sep 24. PMID 19781877
- [Result] Dutton GR, Napolitano MA, Whiteley JA, Marcus BH. Is physical activity a gateway behavior for diet? Findings from a physical activity trial. Prev Med. 2008 Mar;46(3):216-21. doi: 10.1016/j.ypmed.2007.12.012. Epub 2008 Jan 29. PMID 18234327